CLINICAL TRIAL: NCT04091685
Title: Added Value of Tc99m Dimercaptosuccinic Acid SPECT Versus Planar Imaging in Detection of Renal Cortical Defects
Brief Title: D Tc 99m Dimercaptosuccinic Acid SPECT Versus Planar
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Sayed Mohamed, Resident doctor, Assiut University
Other Study IDs: DSVP
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Dimercaptosuccinic Acid SPECT and Planar
MeSH Terms: interventions — Radionuclide Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Gamma camera imaging — Use gamma camera in detection of renal cortical defects

SUMMARY:
Knowing what will DMSA spect add to the DMSA planar in detection in renal cortical defects

ELIGIBILITY:
Inclusion Criteria:

* patient with history of peylo nephritis.

Exclusion Criteria:

* pregnant women

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient with history of peylo nephritis ,malrotated kidney ,ectopic kidney with no age limitation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Comparison between DMSA spect and planar imaging | Baseline
  Analysis of DMSA spect and planar imaging to clarify early renal cortical defects

SECONDARY OUTCOMES:
Clarify added value of DMSA spect over planar | Baseline
  Know if DMSA spect is necessary?

IPD SHARING:
Plan to Share IPD: Undecided